CLINICAL TRIAL: NCT07304388
Title: Systemic Chemotherapy, Lenvatinib and Toripalimab With or Without Hepatic Arterial Infusion In Advanced Intrahepatic Cholangiocarcinoma: A Prospective, Randomized, Two-Cohort, Phase II Study.
Brief Title: HAIC Plus Systemic Chemotherapy, Lenvatinib and Toripalimab in Advanced ICC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IA3GM-II
Record Dates: First submitted 2025-12-11; First posted 2025-12-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc)
Keywords: HAIC; GemOx; combined therapy; lenvatinib; immunotherapy
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm: Hepatic arterial infusion plus systemic chemotherapy, lenvatinib and toripalimab (Experimental)
  Interventions: Procedure: hepatic arterial infusion chemotherapy (HAIC)
- Control arm: Gemox plus lenvatinib and toripalimab (Active Comparator)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Procedure: hepatic arterial infusion chemotherapy (HAIC) — Hepatic arterial infusion chemotherapy:
  oxaliplatin 85mg/m2 via HAIC pump for 3 hours on day 1; Q3W Drug: Gemcitabine
  1g/m2 intravenously on day 1 and day 8 of a 3 weeks cycle Drug: Lenvatinib 12 mg (or 8 mg) once daily (QD) oral dosing Drug: Toripalimab 240 mg iv.drip Q3W
  Arms: Experimental arm: Hepatic arterial infusion plus systemic chemotherapy, lenvatinib and toripalimab
Drug: Chemotherapy — Systemic chemotherapy of GemOx regimen:
  oxaliplatin 85mg/m2 and gemcitabine 1g/m2 intravenously on day 1, and gemcitabine 1g/m2 intravenously on day 8 of a 3 weeks cycle.
  Drug: Lenvatinib 12 mg (or 8 mg) once daily (QD) oral dosing Drug: Toripalimab 240 mg iv.drip Q3W
  Arms: Control arm: Gemox plus lenvatinib and toripalimab

SUMMARY:
Prognosis for unresectable intrahepatic cholangiocarcinoma (ICC) remains poor. Treatment combination known as Gemox (systemic chemotherapy of gemcitabine and oxaliplatin), along with lenvatinib and toripalimab, has shown favor results for ICC patients. However, Hepatic Arterial Infusion Chemotherapy (HAIC), which delivers chemotherapy directly to the liver, has also demonstrated benefits in controlling the cancer locally and improving survival for patients with ICC.

Based on these promising approaches, this study aims to find out if adding HAIC to the systemic chemotherapy-based treatment can help extending patients survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven ICC with locally advanced or metastatic disease deemed unresectable by multidisciplinary evaluation; At least one measurable disease according to the Response Evaluation Criteria in Solid Tumors（RECIST v1.1）; Child-Pugh class A or B; ECOG performance status 0-1; Adequate bone marrow function（white blood cell count ≥2,000cells/mm3, hemoglobin > 9.0 g/dL, Platelet count ≥75,000/mm3）; Adequate hepatic and renal function (albumin ≥ 30 g/L, total bilirubin < 3 times the upper limit of normal, aspartate and alanine transaminases < 5 times the upper limit of normal, creatinine clearance rate of ≤ 1.5 times the upper limit of the normal) and coagulation function（PT < 18s, INR < 1.26）; written informed consent.

Exclusion Criteria:

* Life expectancy less than 2 months; concurrent other malignancy; Prior anticancer therapy (including chemotherapy, radiotherapy, surgery, or interventional treatments); Known allergy to chemotherapy drugs, lenvatinib or PD-(L)1 inhibitors; Patients with uncontrolled comorbidities, active infections; pregnancy or lactation; Refuse to comply with study and/or follow-up procedures; Gastrointestinal bleeding of any grade within 4 weeks prior to the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
6-months PFS | 6 months
  6-months Progression-Free Survival Rate (6-months PFS rate) is defined as the proportion of patients who remain alive and free from disease progression (as assessed by RECIST v1.1) at 6 months from the initiation of study randomization.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 18 months
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on RECIST. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference to the baseline sum of the diameters of target lesions.
Overall Survival (OS) | 18 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.
Progression Free Survival (PFS) | 18 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first.
Adverse Events | 30 days
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China